CLINICAL TRIAL: NCT04847674
Title: A Phase 2, Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Assess the Safety, Efficacy and Pharmacodynamics of TEV 53275 Administered Subcutaneously in Adult Patients With Persistent Eosinophilic Asthma
Brief Title: A Study to Test if TEV-53275 is Effective in Relieving Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped for strategic reasons
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV53275-AS-20033; 2021-001439-22 (EudraCT Number)
Record Dates: First submitted 2021-04-05; First posted 2021-04-19 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Persistent; Eosinophilic; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TEV-53275 Dose A (Experimental)
  Interventions: Drug: TEV-53275 Dose A
- TEV-53275 Dose B (Experimental)
  Interventions: Drug: TEV-53275 Dose B
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-53275 Dose A — subcutaneous (sc) injection
  Arms: TEV-53275 Dose A
Drug: TEV-53275 Dose B — subcutaneous (sc) injection
  Arms: TEV-53275 Dose B
Drug: Placebo — Matching subcutaneous (sc) placebo injection
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of TEV-53275 administered subcutaneously (sc) in adult participants with persistent asthma and an eosinophilic phenotype compared to placebo. A secondary objective is to evaluate the efficacy of TEV-53275 compared to placebo assessed by lung function, asthma symptoms, rescue medication use, and quality of life measures. Another secondary objective is to evaluate the safety and tolerability of TEV-53275 administered sc in adult participants with persistent asthma and an eosinophilic phenotype compared with placebo, and lastly, to evaluate the immunogenicity of TEV-53275 administered sc in adult participants with persistent asthma and an eosinophilic phenotype.

DETAILED DESCRIPTION:
The planned study duration is approximately 16 months.

The total duration of study participation is approximately 34 weeks including up to a 2-week screening period, a 2-week run-in period, a 16-week treatment period, and a follow-up visit 14 weeks after the final treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* The participant is an adult female or male ≥18 years of age. Note: Age requirements are as specified or allowed by local regulations.
* The participant has a diagnosis of asthma for at least 6 months and has been stable without exacerbation or change in medications for at least 1 month..
* Current Asthma Therapy: The participant has been maintained for at least 1 month on stable doses of:

  * medium or high dose inhaled corticosteroids (ICS)±another controller.
  * any fixed dose combination ICS (low, medium, or high) with long-acting beta agonist (LABA)±another controller.
* Women of non-childbearing potential, or congenitally sterile, or 1-year postmenopausal. Women of childbearing potential must have a negative β-human chorionic gonadotropin (β-HCG) test result and practice a highly effective method of birth control prior to investigational medicinal product (IMP) administration and 30 weeks after the dose of IMP.
* The participant, as judged by the investigator, is able to continue their current asthma maintenance medications throughout the study.

NOTE- Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* Life threatening asthma, defined as a history of asthma episode(s) requiring intubation and/or associated hypercapnea, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s).
* The participant has a suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the screening period. Note: Participants who develop an upper respiratory infection/lower respiratory infection (URI/LRI) during the run-in period may rescreen 2 weeks after symptoms resolve and undergo coronavirus disease 2019 (COVID-19) testing.
* Participants with a confirmed infection with COVID-19 within 3 months prior to the screening visit.
* The participant has an eosinophilic condition including hypereosinophilic syndrome, eosinophilic pneumonia, eosinophilic granulomatosis with polyangiitis (EGPA [Churg Strauss syndrome]), or allergic bronchopulmonary aspergillosis.
* The participant has an active helminthic or parasitic infection currently or within the last 6 months.
* The participant has a history of malignancy other than fully resected basal cell carcinoma of the skin.
* The participant has any clinically significant, uncontrolled medical or psychiatric condition (treated or untreated) that would interfere with the study schedule or procedures, interpretation of efficacy results, or compromise the participant's safety.
* The participant has known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies (Ab), or human immunodeficiency virus (HIV) Types 1 or 2 Ab (according to 4th generation serology testing).
* The participant is a pregnant or lactating woman, or plans to become pregnant during the study.
* The participant has previously participated in a study with TEV-53275.
* The participant has participated in another study of an IMP (or a medical device) within the previous 30 days or is currently participating in another study of an IMP (or a medical device).
* The participant has been treated with a monoclonal antibody used to treat asthma or other inflammatory conditions within the washout period (5 half-lives), has demonstrated hypersensitivity or anaphylaxis to a monoclonal antibody (Appendix G),or is currently using or has used a systemic immunosuppressive medication within the last 6 months. NOTE: Prior depemokimab exposure is prohibited without exception.
* The participant has a history of chronic alcohol or drug abuse within the previous 2 years.
* The participant currently smokes or has a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes [20 cigarettes]/day for 1 year), OR the participant used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco), OR the participant has smoked marijuana within 1 month, OR the participant has a history of "vaping" tobacco, marijuana, or any other substance within 24 months.
* Vulnerable participants (eg, people kept in detention).

NOTE- Additional criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (82):
- United States (77):
  - Teva Investigational Site 15188, Hoover, Alabama
  - Teva Investigational Site 15174, Peoria, Arizona
  - Teva Investigational Site 15202, Phoenix, Arizona
  - Teva Investigational Site 15205, Tucson, Arizona
  - Teva Investigational Site 15178, Bakersfield, California
  - Teva Investigational Site 15196, Bakersfield, California
  - Teva Investigational Site 15176, Encinitas, California
  - Teva Investigational Site 15156, Huntington Beach, California
  - Teva Investigational Site 15209, Inglewood, California
  - Teva Investigational Site 15194, Los Angeles, California
  - Teva Investigational Site 15143, Los Angeles, California
  - Teva Investigational Site 15212, Los Angeles, California
  - Teva Investigational Site 15151, Mission Viejo, California
  - Teva Investigational Site 15210, North Hollywood, California
  - Teva Investigational Site 15136, San Jose, California
  - Teva Investigational Site 15157, Stockton, California
  - Teva Investigational Site 15158, Upland, California
  - Teva Investigational Site 15167, Walnut Creek, California
  - Teva Investigational Site 15133, Westminster, California
  - Teva Investigational Site 15166, Colorado Springs, Colorado
  - Teva Investigational Site 15200, Lafayette, Colorado
  - Teva Investigational Site 15139, Wheat Ridge, Colorado
  - Teva Investigational Site 15182, Boynton Beach, Florida
  - Teva Investigational Site 15147, Hialeah, Florida
  - Teva Investigational Site 15134, Hialeah, Florida
  - Teva Investigational Site 15152, Leesburg, Florida
  - Teva Investigational Site 15149, Miami, Florida
  - Teva Investigational Site 15211, Miami, Florida
  - Teva Investigational Site 15206, Miami, Florida
  - Teva Investigational Site 15215, Miami, Florida
  - Teva Investigational Site 15141, Miami, Florida
  - Teva Investigational Site 15169, Miami Lakes, Florida
  - Teva Investigational Site 15170, North Palm Beach, Florida
  - Teva Investigational Site 15130, Orlando, Florida
  - Teva Investigational Site 15140, Tallahassee, Florida
  - Teva Investigational Site 15132, Tampa, Florida
  - Teva Investigational Site 15135, Sugar Hill, Georgia
  - Teva Investigational Site 15183, Normal, Illinois
  - Teva Investigational Site 15198, Overland Park, Kansas
  - Teva Investigational Site 15187, Zachary, Louisiana
  - Teva Investigational Site 15148, Baltimore, Maryland
  - Teva Investigational Site 15190, North Dartmouth, Massachusetts
  - Teva Investigational Site 15175, Columbia, Missouri
  - Teva Investigational Site 15145, Rolla, Missouri
  - Teva Investigational Site 15144, St Louis, Missouri
  - Teva Investigational Site 15137, Bellevue, Nebraska
  - Teva Investigational Site 15164, Skillman, New Jersey
  - Teva Investigational Site 15165, The Bronx, New York
  - Teva Investigational Site 15181, Charlotte, North Carolina
  - Teva Investigational Site 15179, Elizabeth City, North Carolina
  - Teva Investigational Site 15193, Greensboro, North Carolina
  - Teva Investigational Site 15153, Monroe, North Carolina
  - Teva Investigational Site 15168, Raleigh, North Carolina
  - Teva Investigational Site 15173, Cincinnati, Ohio
  - Teva Investigational Site 15131, Toledo, Ohio
  - Teva Investigational Site 15201, Edmond, Oklahoma
  - Teva Investigational Site 15204, Tulsa, Oklahoma
  - Teva Investigational Site 15180, Medford, Oregon
  - Teva Investigational Site 15172, Portland, Oregon
  - Teva Investigational Site 15192, Jenkintown, Pennsylvania
  - Teva Investigational Site 15185, Pittsburgh, Pennsylvania
  - Teva Investigational Site 15161, Clinton, South Carolina
  - Teva Investigational Site 15159, Rock Hill, South Carolina
  - Teva Investigational Site 15162, Austin, Texas
  - Teva Investigational Site 15138, Dallas, Texas
  - Teva Investigational Site 15154, Dallas, Texas
  - Teva Investigational Site 15171, Denton, Texas
  - Teva Investigational Site 15155, El Paso, Texas
  - Teva Investigational Site 15189, Houston, Texas
  - Teva Investigational Site 15184, Houston, Texas
  - Teva Investigational Site 15199, Houston, Texas
  - Teva Investigational Site 15191, Houston, Texas
  - Teva Investigational Site 15160, McKinney, Texas
  - Teva Investigational Site 15197, San Antonio, Texas
  - Teva Investigational Site 15195, Williamsburg, Virginia
  - Teva Investigational Site 15150, Bellingham, Washington
  - Teva Investigational Site 15142, Greenfield, Wisconsin
- Canada (5):
  - Teva Investigational Site 11218, Sherwood Park, Alberta
  - Teva Investigational Site 11212, Ajax, Ontario
  - Teva Investigational Site 11211, Toronto, Ontario
  - Teva Investigational Site 11213, Montreal, Quebec
  - Teva Investigational Site 11214, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to TEV-53275 subcutaneously (SC) at baseline (Day 0).
- TEV-53275 Dose A: Participants received TEV-53275 Dose A SC at baseline (Day 0).
- TEV-53275 Dose B: Participants received TEV-53275 Dose B SC at baseline (Day 0).
Period: Overall Study
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Started | 32 | 33 | 32
Received at Least 1 Dose of Study Drug as Randomized | 31 | 33 | 32
Modified Intent-to-treat (mITT) Analysis Set (All randomized participants who received at least a partial dose of study drug.) | 31 | 33 | 32
Safety Analysis Set (All randomized participants who received at least 1 dose of study drug. In this set, data were summarized based upon the treatment actually received regardless of the assigned treatment.) | 31 | 34 (One participant was randomized to TEV-53275 Dose B but received TEV-53275 Dose A. Therefore, the participant was included in the TEV-53275 Dose A arm for the Safety Analysis Set.) | 31
Completed | 11 | 12 | 10
Not Completed | 21 | 21 | 22
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Other than specified | 21 | 20 | 20

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: Participants received placebo matched to TEV-53275 SC at baseline (Day 0).
- Total: Total of all reporting groups
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B | Total
Number analyzed (Participants) | 32 | 33 | 32 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.94) | 51.2 (13.79) | 53.2 (15.05) | 51.9 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 19 | 60
  Male | 9 | 15 | 13 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 5 | 18
  Not Hispanic or Latino | 28 | 24 | 27 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 1 | 13
  White | 25 | 25 | 29 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] — Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug.
  liters
    number analyzed (Participants) | 31 | 33 | 32 | 96
    (all) | 1.938 (0.5931) | 1.957 (0.6961) | 2.064 (0.7411) | 1.986 (0.6757)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic-based Standardized Baseline-adjusted Morning Trough (Pre-bronchodilator) FEV1 at Week 12
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. Least square (LS) mean and standard error (SE) were calculated using a mixed model for repeated measures (MMRM).
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 24 | 26 | 27
liters | 0.152 (0.0746) | 0.125 (0.0724) | 0.140 (0.0718)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using an MMRM with treatment group, week, randomization factors, and treatment group by week interaction as fixed effects, and baseline FEV1 as a covariate; Test type: Other; p = 0.7914, Mixed Models Analysis; LS mean difference = -0.027, 95% CI 2-sided [-0.2276 to 0.1740]
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9115, Mixed Models Analysis; LS mean difference = -0.011, 95% CI 2-sided [-0.2126 to 0.1900]

2. Secondary Outcome: Number of Participants With Well-controlled Asthma Status (Yes Versus No) at Weeks 12 and 16
Description: The weekly asthma control status (Yes or No) is the derived asthma control composite score based on the following criteria:
  1. Two or more of the following criteria were fulfilled:
  * ≤2 days with a daily asthma symptom score >1; - ≤2 days of albuterol/salbutamol used as rescue medication up to a maximum of 4 occasions per week (multiple occasions per day are counted as separate occasions); - morning FEV1 ≥80% predicted for each day (by handheld device) and 2. Both of the following criteria were fulfilled:
  * no night-time awakenings due to asthma; - no use of asthma maintenance medications.
  The asthma control status in each weekly analysis window was Yes if the conditions 1 and 2 above were met, No otherwise.
Time Frame: Weeks 12 and 16
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed = participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 23 | 26 | 27
Participants
  Well-controlled asthma status at Week 12: Yes | 6 | 11 | 6
  Well-controlled asthma status at Week 12: No | 17 | 15 | 21
  Well-controlled asthma status at Week 16: number analyzed (Participants) | 23 | 24 | 26
  Well-controlled asthma status at Week 16: Yes | 6 | 12 | 6
  Well-controlled asthma status at Week 16: No | 17 | 12 | 20

3. Secondary Outcome: Change From Baseline in the Weekly Average of Daily Morning Trough (Pre-Rescue Bronchodilator) FEV1 Over 12 Weeks From Week 1 Through 12 and Over 16 Weeks From Week 1 Through 16
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by a handheld device. The post-baseline analysis window for over 12 weeks was from the first day of study drug up to Day 84. The post-baseline analysis window for over 16 weeks was from the first day of study drug up to Day 112. The daily average of the efficacy data with each weekly analysis window was calculated based on non-missing e-diary as follow: Summation of FEV1 during an analysis window/Number of days with nonmissing data in the analysis window. LS mean and SE was calculated using an MMRM.
Time Frame: Baseline, up to Week 12, up to Week 16
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 33 | 32
liters
  Change over 12 weeks | 0.007 (0.0373) | 0.034 (0.0365) | 0.034 (0.0362)
  Change over 16 weeks | 0.009 (0.0378) | 0.036 (0.0369) | 0.032 (0.0367)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6001, Mixed Models Analysis; LS mean difference = 0.026, 95% CI 2-sided [-0.0733 to 0.1261] — Change from baseline in FEV1 over 12 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5922, Mixed Models Analysis; LS mean difference = 0.027, 95% CI 2-sided [-0.0732 to 0.1276] — Change from baseline in FEV1 over 12 weeks: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6017, Mixed Models Analysis; LS mean difference = 0.027, 95% CI 2-sided [-0.0744 to 0.1277] — Change from baseline in FEV1 over 16 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6664, Mixed Models Analysis; LS mean difference = 0.022, 95% CI 2-sided [-0.0796 to 0.1239] — Change from baseline in FEV1 over 16 weeks: TEV-53275 Dose B versus Placebo

4. Secondary Outcome: Change From Baseline in Weekly Average of Rescue Medication Use Over 12 Weeks From Week 1 Through 12 and Over 16 Weeks From Week 1 Through 16
Description: The number of times asthma rescue medication (number of inhalations/puffs) was used was assessed (for example, by reviewing the electronic diary or if required due to missing data in the diary, by site tracking of the inhalation counter on the inhaler). Rescue medication included albuterol sulfate inhalation powder (albuterol eMDPI) or equivalent albuterol/salbutamol. The post-baseline analysis window for over 12 weeks was from the first day of study drug up to Day 84. The post-baseline analysis window for over 16 weeks was from the first day of study drug up to Day 112. The daily average of the efficacy data with each weekly analysis window was calculated based on non-missing e-diary as follow: Summation of rescue medication uses during an analysis window/Number of days with nonmissing data in the analysis window. LS mean and SE were calculated using Wilcoxon rank-sum test stratified on randomization stratification factors.
Time Frame: Baseline, up to Week 12, up to Week 16
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug.
Measure: Mean (Standard Deviation); unit: number of inhalations/week
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 33 | 32
number of inhalations/week
  Change in weekly average rescue medication use over 12 weeks | -3.7 (9.21) | -3.4 (5.86) | -2.9 (8.55)
  Change in weekly average rescue medication use over 16 weeks | -4.2 (9.30) | -3.5 (5.81) | -3.0 (8.66)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using Wilcoxon rank-sum test stratified on randomization stratification factors; Test type: Other; p = 0.7261, Wilcoxon (Mann-Whitney); Hodges-Lehmann (HL) estimator = 0.4, 95% CI 2-sided [-2.33 to 3.31] — Change from baseline in weekly average of rescue medication use over 12 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; Analysis was performed using Wilcoxon rank-sum test stratified on randomization stratification factors; Test type: Other; p = 0.7650, Wilcoxon (Mann-Whitney); HL estimator = -0.5, 95% CI 2-sided [-3.56 to 3.32] — Change from baseline in weekly average of rescue medication use over 12 weeks: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using Wilcoxon rank-sum test stratified on randomization stratification factors; Test type: Other; p = 0.7942, Wilcoxon (Mann-Whitney); HL estimator = 0.2, 95% CI 2-sided [-2.44 to 3.04] — Change from baseline in weekly average of rescue medication use over 16 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; Analysis was performed using Wilcoxon rank-sum test stratified on randomization stratification factors; Test type: Other; p = 0.6147, Wilcoxon (Mann-Whitney); HL estimator = -0.8, 95% CI 2-sided [-3.81 to 2.55] — Change from baseline in weekly average of rescue medication use over 16 weeks: TEV-53275 Dose B versus Placebo

5. Secondary Outcome: Change From Baseline in Weekly Percentage of Asthma Control Days (No Symptoms and No Rescue Medication Use) Over 12 Weeks From Week 1 Through 12 and Over 16 Weeks From Week 1 Through 16
Description: An asthma control day was defined as a day on which the participant used 0 puffs of inhaled short-acting β-adrenergic agonist (SABA), had no night-time awakenings, and experienced no asthma exacerbations. The post-baseline analysis window for over 12 weeks was from the first day of study drug up to Day 84. The post-baseline analysis window for over 16 weeks was from the first day of study drug up to Day 112. Percentage of asthma control days in each analysis window was calculated as follow: Summation of asthma control days in an analysis window/Number of days with nonmissing data in the analysis window * 100.
Time Frame: Baseline, up to Week 12, up to Week 16
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of days/week
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 33 | 32
percentage of days/week
  Change in weekly percentage of asthma control days over 12 weeks | 23.21 (36.645) | 21.51 (23.907) | 12.71 (27.024)
  Change in weekly percentage of asthma control days over 16 weeks | 24.28 (36.557) | 23.23 (25.585) | 13.57 (28.148)

6. Secondary Outcome: Change From Baseline in Clinic-based Standardized Baseline-adjusted Morning Trough (Pre-bronchodilator) FEV1 at Week 16
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer. LS mean and SE were calculated using an MMRM.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 23 | 24 | 26
liters | 0.175 (0.0787) | 0.092 (0.0771) | 0.086 (0.0754)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4394, Mixed Models Analysis; LS mean difference = -0.083, 95% CI 2-sided [-0.2971 to 0.1301]
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4051, Mixed Models Analysis; LS mean difference = -0.089, 95% CI 2-sided [-0.3020 to 0.1231]

7. Secondary Outcome: Number of Participants Who Achieved Clinic-based FEV1 ≥80% Predicted at Weeks 12 and 16
Description: The percent of predicted FEV1 (the volume of air exhaled in the first second of a forced expiration) was measured by handheld device.
Time Frame: Weeks 12 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 21 | 24 | 24
Participants
  Week 12 | 7 | 7 | 8
  Week 16: number analyzed (Participants) | 20 | 22 | 23
  Week 16 | 6 | 4 | 5

8. Secondary Outcome: Number of Participants Who Achieved Forced Expiratory Flow at 25% to 75% of Forced Expiratory Volume (FVC) (FEF25-75) ≥70% Predicted at Weeks 12 and 16
Description: The FVC is the volume of air that can be forcibly blown out after full inspiration. FVC results in this study were presented as the forced expiratory flow at 25% to 75% of FVC.
Time Frame: Weeks 12 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 22 | 24 | 25
Participants
  Week 12 | 2 | 3 | 1
  Week 16: number analyzed (Participants) | 21 | 23 | 24
  Week 16 | 2 | 2 | 2

9. Secondary Outcome: Change From Baseline in FEF25-75 Over 12 Weeks From Week 1 Through 12 and Over 16 Weeks From Week 1 Through 16
Description: The FVC is the volume of air that can be forcibly blown out after full inspiration. FVC results in this study were presented as the forced expiratory flow at 25% to 75% of FVC. The post-baseline analysis window for over 12 weeks was from the first day of study drug up to Day 84. The post-baseline analysis window for over 16 weeks was from the first day of study drug up to Day 112. The daily average of the efficacy data with each weekly analysis window was calculated based on non-missing e-diary as follow: Summation of FEF25-75 during an analysis window/Number of days with nonmissing data in the analysis window. LS mean and SE were calculated using an MMRM.
Time Frame: Baseline, up to Week 12, up to Week 16
Population: The mITT analysis set included all randomized participants who received at least a partial dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 33 | 32
liters/second
  Change in FEF25-75 over 12 weeks | 0.086 (0.0742) | 0.179 (0.0734) | 0.119 (0.0721)
  Change in FEF25-75 over 16 weeks | 0.098 (0.0772) | 0.185 (0.0763) | 0.108 (0.0749)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using an MMRM with treatment group, week, randomization factors, and treatment group by week interaction as fixed effects, and baseline FEF25-75 as a covariate; Test type: Other; p = 0.3485, Mixed Models Analysis; LS mean difference = 0.093, 95% CI 2-sided [-0.1031 to 0.2893] — Change from baseline in FEF25-75 over 12 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.7432, Mixed Models Analysis; LS mean difference = 0.033, 95% CI 2-sided [-0.1644 to 0.2296] — Change from baseline in FEF25-75 over 12 weeks: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.4014, Mixed Models Analysis; LS mean difference = 0.087, 95% CI 2-sided [-0.1180 to 0.2920] — Change from baseline in FEF25-75 over 16 weeks: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.9259, Mixed Models Analysis; LS mean difference = 0.010, 95% CI 2-sided [-0.1960 to 0.2153] — Change from baseline in FEF25-75 over 16 weeks: TEV-53275 Dose B versus Placebo

10. Secondary Outcome: Time to First Clinical Asthma Exacerbation (CAE)
Description: The time (days) to the first CAE was the interval from the randomization to the occurrence of the first CAE. A CAE was defined as worsening asthma requiring treatment with a systemic corticosteroid for at least 3 days, emergency room visit resulting in systemic corticosteroid treatment, or hospitalization due to asthma. Worsening asthma included new or increased symptoms or signs that either worried the participant or were related to an asthma-specific alert (if available through the electronic diary/handheld spirometer) and required the addition of maintenance medications (other than systemic corticosteroids) to control the participant's asthma symptoms based on the investigator's judgment.
Time Frame: Baseline up to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 2 | 3 | 2
days | 54.5 (36.06) | 77.0 (47.82) | 87.0 (36.77)

11. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-6) Score at Weeks 12 and 16
Description: The ACQ-6 is a validated 6-item asthma assessment tool that has been widely used. Six questions are self-assessments (completed by the participant), 5 questions assessing asthma symptoms: night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and 1 question for short-acting bronchodilator use. Each item on the ACQ has a possible score ranging from 0 (no impairment) to 6 (maximum impairment), and the total score is the mean of all responses. The total score ranging from 0 (totally controlled) to 6 (severely uncontrolled) with higher scores indicating maximum impairment.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 24 | 26 | 27
units on a scale
  Change in ACQ-6 score at Week 12 | -1.1 (0.16) | -1.1 (0.16) | -1.0 (0.15)
  Change in ACQ-6 score at Week 16: number analyzed (Participants) | 23 | 25 | 26
  Change in ACQ-6 score at Week 16 | -1.0 (0.16) | -1.1 (0.16) | -1.0 (0.16)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using an MMRM with treatment group, week, randomization factors, and treatment group by week interaction as fixed effects, and baseline ACQ-6 as a covariate; Test type: Other; p = 0.9829, Mixed Models Analysis; LS mean difference = 0.0, 95% CI 2-sided [-0.43 to 0.42] — Change from baseline in ACQ-6 at Week 12: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 11, analysis 1]; Test type: Other; p = 0.6302, Mixed Models Analysis; LS mean difference = 0.1, 95% CI 2-sided [-0.32 to 0.52] — Change from baseline in ACQ-6 at Week 12: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 11, analysis 1]; Test type: Other; p = 0.6707, Mixed Models Analysis; LS mean difference = -0.1, 95% CI 2-sided [-0.54 to 0.35] — Change from baseline in ACQ-6 at Week 16: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 11, analysis 1]; Test type: Other; p = 0.9940, Mixed Models Analysis; LS mean difference = 0.0, 95% CI 2-sided [-0.44 to 0.43] — Change from baseline in ACQ-6 at Week 16: TEV-53275 Dose B versus Placebo

12. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Score at Weeks 12 and 16
Description: The Asthma Control Test (ACT) is a participant self-administered tool for identifying those with poorly controlled asthma comprising 5 items, with 4-week recall (on symptoms and daily functioning). It assesses the frequency of shortness of breath and general asthma symptoms, the use of rescue medications, the effect of asthma on daily functioning, and the overall self-assessment of asthma control measured on a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). Total scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 24 | 26 | 27
units on a scale
  Change at Week 12 | 4.8 (0.75) | 4.1 (0.73) | 3.6 (0.70)
  Change at Week 16: number analyzed (Participants) | 23 | 25 | 26
  Change at Week 16 | 4.6 (0.72) | 4.0 (0.71) | 3.7 (0.68)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using an MMRM with treatment group, week, randomization factors, and treatment group by week interaction as fixed effects, and baseline ACT as a covariate; Test type: Other; p = 0.4683, Mixed Models Analysis; LS mean difference = -0.7, 95% CI 2-sided [-2.71 to 1.26] — Change from baseline in ACT at Week 12: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.2239, Mixed Models Analysis; LS mean difference = -1.2, 95% CI 2-sided [-3.16 to 0.75] — Change from baseline in ACT at Week 12: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.5389, Mixed Models Analysis; LS mean difference = -0.6, 95% CI 2-sided [-2.51 to 1.32] — Change from baseline in ACT at Week 16: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 12, analysis 1]; Test type: Other; p = 0.3564, Mixed Models Analysis; LS mean difference = -0.9, 95% CI 2-sided [-2.75 to 1.00] — Change from baseline in ACT at Week 16: TEV-53275 Dose B versus Placebo

13. Secondary Outcome: Change From Baseline in Standardized Asthma Quality of Life Questionnaire (AQLQ[S]) Overall Score at Weeks 12 and 16
Description: The AQLQ[S] (participants ≥18 years of age version) was self-administered by participants. The questionnaire is a tool to measure the impact of asthma on a participant's quality of life (physical, emotional, social, and occupational). The aim of the questionnaire is to evaluate the problems that were most troublesome to participants in their day to day lives. The questionnaire contains 32 items with a 2-week recall period and used a 7-point Likert scale (7=not impaired at all to 1=severely impaired). The overall AQLQ score was the mean of the responses to each of the 32 questions and ranged from 1 (severely impaired) to 7 (not impaired at all) with higher scores indicating better quality of life.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 32 | 32
units on a scale
  Change at Week 12 | 1.0 (0.17) | 0.8 (0.17) | 0.8 (0.16)
  Change at Week 16: number analyzed (Participants) | 23 | 25 | 26
  Change at Week 16 | 0.9 (0.18) | 0.7 (0.18) | 0.8 (0.17)
Statistical Analysis 1: Comparison: Placebo vs TEV-53275 Dose A; Analysis was performed using an MMRM with treatment group, week, randomization factors, and treatment group by week interaction as fixed effects, and baseline AQLQ as a covariate; Test type: Other; p = 0.4436, Mixed Models Analysis; LS mean difference = -0.2, 95% CI 2-sided [-0.62 to 0.27] — Change from baseline in AQLQT at Week 12: TEV-53275 Dose A versus Placebo
Statistical Analysis 2: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.5970, Mixed Models Analysis; LS mean difference = -0.1, 95% CI 2-sided [-0.56 to 0.32] — Change from baseline in AQLQT at Week 12: TEV-53275 Dose B versus Placebo
Statistical Analysis 3: Comparison: Placebo vs TEV-53275 Dose A; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.3769, Mixed Models Analysis; LS mean difference = -0.2, 95% CI 2-sided [-0.68 to 0.26] — Change from baseline in AQLQT at Week 16: TEV-53275 Dose A versus Placebo
Statistical Analysis 4: Comparison: Placebo vs TEV-53275 Dose B; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.4595, Mixed Models Analysis; LS mean difference = -0.2, 95% CI 2-sided [-0.64 to 0.29] — Change from baseline in AQLQT at Week 16: TEV-53275 Dose B versus Placebo

14. Secondary Outcome: Number of Participants Who Achieved FEV1:FVC Ratio ≥0.80 at Weeks 12 and 16
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration. FVC is the volume of air that can be forcibly blown out after full inspiration.
Time Frame: Weeks 12 and 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 20 | 22 | 26
Participants
  Week 12 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 19 | 21 | 25
  Week 16 | 0 | 0 | 2

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that occurred after the first dose of study drug was administered through the end of the study. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 30
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. In this set, data were summarized based upon the treatment actually received regardless of the assigned treatment. One participant was randomized to TEV-53275 Dose B but received TEV-53275 Dose A. Therefore, the participant was included in the TEV-53275 Dose A arm for the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 11 | 22 | 14

16. Secondary Outcome: Number of Participants Who Received at Least 1 Concomitant Asthma Medication
Description: Concomitant asthma medications included Antihistamines for systemic use (Cetirizine); Corticosteroids for systemic use (Prednisone, Methylprednisolone); and Drugs for obstructive airway diseases (Salbutamol, Fluticasone etc.).
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 31 | 34 | 31

17. Secondary Outcome: Number of Participants Developing Antidrug Antibodies (ADAs) Throughout the Study
Description: A participant was classified as having a treatment-emergent ADA response if either of the following were true: - The participant had a positive sample at any of the postdose time points, but not at the predose (baseline) time point; - The participant had a positive sample at predose (baseline) and 1 or more postdose time points, but the titer of a postdose sample(s) was increased by at least 4-fold when comparing it to that of the predose sample.
Time Frame: Baseline up to Week 30
Population: The ADA analysis set (for anti-TEV-53275 antibodies) included those participants treated with TEV-53275 in the safety analysis set. In this set, data were summarized based upon the treatment actually received regardless of the assigned treatment. One participant was randomized to TEV-53275 Dose B but received TEV-53275 Dose A. Therefore, the participant was included in the TEV-53275 Dose A arm for the ADA Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 34 | 31
Participants | 1 | 0

18. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Serum Chemistry Value
Description: Potentially clinically significant serum chemistry abnormalities included: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase, Gamma-glutamyl transpeptidase (GGT), Lactate dehydrogenase (LDH), and Creatinine phosphokinase each ≥3 * upper limit of normal (ULN); Blood urea nitrogen ≥10.71 millimoles (mmol)/liter (L); Creatinine ≥177 micromoles (μmol)/L; and Bilirubin (total) ≥34.2 μmol /L.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 2 | 3 | 2

19. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Hematology Value
Description: Potentially clinically significant hematological abnormalities included: White blood cells (WBCs) count ≤3.0 *10^9 cells/L or ≥20 * 10^9 cells/L; Hemoglobin ≤95 grams (g)/L in females and ≤115 g/L in males; Hematocrit <0.32 L/L in females and <0.37 L/L in males; Platelet count ≤75 * 10^9 cells/L or ≥700 * 10^9 cells/L; and Absolute neutrophil count (ANC) ≤1 * 10^9 cells/L.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 1 | 2 | 0

20. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Urinalysis Abnormalities
Description: Potentially clinically significant urinalysis abnormalities included: ≥2 unit increase from baseline in urine hemoglobin, ketones, glucose, and total protein.
Time Frame: Baseline up to Week 30
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. In this set, data were summarized based upon the treatment actually received regardless of the assigned treatment. One participant was randomized to TEV-53275 Dose B but received TEV-53275 Dose A. Therefore, the participant was included in the TEV-53275 Dose A arm for the Safety Analysis Set. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 33 | 31
Participants | 4 | 3 | 3

21. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Vital Signs Value
Description: Potentially clinically significant vital signs abnormalities included: Systolic blood pressure (BP): ≤90 millimeters of mercury (mmHg) and decrease from baseline of 20 mm Hg or ≥180 mm Hg and increase from baseline of ≥20 mm Hg; Diastolic BP: ≥105 mmHg and increase from baseline of ≥15 mmHg or ≤50 mmHg and decrease from baseline of ≥15 mmHg; Pulse ≥120 beats per minute (bpm) and increase from baseline of ≥15 bpm or ≤50 bpm and decrease from baseline of ≥15 bpm; Temperature ≥38.3 degrees celsius (ºC) and change from baseline of ≥1.1 ºC; Respiratory rate >24 breaths/min and increase from baseline of ≥10 breaths/min.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 1 | 0 | 0

22. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Electrocardiogram Values
Description: Potentially clinically significant electrocardiogram abnormalities including any one of the following values: QTc interval >450 milliseconds (msec) and QTc interval increases from baseline >30 msec, QTc interval >450 msec and QTc interval increases from baseline >60 msec, QTc interval >500 msec and QTc interval increases from baseline >30 msec, QTc interval >500 msec and QTc interval increases from baseline >60 msec; QRS duration >110 msec and a 25% increase from baseline; and PR interval >200 msec and a 25% increase from baseline.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 0 | 1 | 0

23. Secondary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions included erythema, ecchymosis, induration, tenderness, warmth, and swelling. Number of participants with erythema, ecchymosis, and induration were reported in following categories: Absent; 5 millimeters (mm) to ≤50 mm (mild); >50 mm to ≤100 mm (moderate); and >100 mm (severe). Number of participants with tenderness, warmth, and swelling were reported in following categories: Absent; mild; moderate; and severe.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants
  Erythema: Absent | 27 | 29 | 21
  Erythema: Mild | 4 | 4 | 8
  Erythema: Moderate | 0 | 1 | 2
  Erythema: Severe | 0 | 0 | 0
  Ecchymosis: Absent | 31 | 33 | 30
  Ecchymosis: Mild | 0 | 1 | 1
  Ecchymosis: Moderate | 0 | 0 | 0
  Ecchymosis: Severe | 0 | 0 | 0
  Induration: Absent | 31 | 32 | 29
  Induration: Mild | 0 | 2 | 2
  Induration: Moderate | 0 | 0 | 0
  Induration: Severe | 0 | 0 | 0
  Tenderness: Absent | 26 | 32 | 27
  Tenderness: Mild | 5 | 1 | 2
  Tenderness: Moderate | 0 | 1 | 2
  Tenderness: Severe | 0 | 0 | 0
  Warmth: Absent | 31 | 30 | 30
  Warmth: Mild | 0 | 4 | 1
  Warmth: Moderate | 0 | 0 | 0
  Warmth: Severe | 0 | 0 | 0
  Swelling: Absent | 29 | 30 | 28
  Swelling: Mild | 2 | 3 | 3
  Swelling: Moderate | 0 | 1 | 0
  Swelling: Severe | 0 | 0 | 0

24. Secondary Outcome: Number of Participants Who Did Not Complete the Study Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Number of participants who did not complete the study due to AEs were reported.
Time Frame: Baseline up to Week 30
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
Number analyzed (Participants) | 31 | 34 | 31
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 30
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug. In this set, data were summarized based upon the treatment actually received regardless of the assigned treatment. One participant was randomized to TEV-53275 Dose B but received TEV-53275 Dose A. Therefore, the participant was included in the TEV-53275 Dose A arm for the Safety Analysis Set.
Arm/Group | Placebo | TEV-53275 Dose A | TEV-53275 Dose B
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/34 | 1/31
Other Adverse Events (participants affected / at risk) | 5/31 | 10/34 | 1/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | TEV-53275 Dose A (N=34) | TEV-53275 Dose B (N=31)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | TEV-53275 Dose A (N=34) | TEV-53275 Dose B (N=31)
COVID-19 (Infections and infestations) | 3 (4) | 6 (6) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT04847674/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT04847674/SAP_001.pdf